CLINICAL TRIAL: NCT04983407
Title: A Phase 1b/2 Randomized Study of AVB-S6-500 Plus Nab-paclitaxel and Gemcitabine in Patients With Locally Advanced or Metastatic Pancreatic Adenocarcinoma
Brief Title: Safety and Efficacy Study of AVB-S6-500 (Batiraxcept) in Patients With Advanced Pancreatic Adenocarcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to business reasons
Sponsor: Aravive, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVB500-PC-005
Record Dates: First submitted 2021-07-08; First posted 2021-07-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: locally advanced; recurrent; metastatic; pancreatic; exocrine; pancreas; adenocarcinoma
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis; Adenocarcinoma | interventions — Taxes; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1b: batiraxcept+ nab-paclitaxel and gemcitabine (Experimental): Up to three dose levels of bactiraxcept plus nab-paclitaxel and gemcitabine
  Interventions: Drug: batiraxcept; Drug: Nab paclitaxel; Drug: Gemcitabine
- Phase 2: batiraxcept+ nab-paclitaxel and gemcitabine (Experimental)
  Interventions: Drug: batiraxcept; Drug: Nab paclitaxel; Drug: Gemcitabine
- Phase 2: nab-paclitaxel and gemcitabine alone (Active Comparator)
  Interventions: Drug: Nab paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: batiraxcept — Batiraxcept is experimental drug
  Other Names: AVB-S6-500
  Arms: Phase 1b: batiraxcept+ nab-paclitaxel and gemcitabine; Phase 2: batiraxcept+ nab-paclitaxel and gemcitabine
Drug: Nab paclitaxel — Nab paclitaxel is active comparator
  Other Names: Abraxane
Drug: Gemcitabine — Gemcitabine is active comparator

SUMMARY:
This is a Phase 1b/2 study of batiraxcept (AVB-S6-500) designed to evaluate the safety and efficacy of batiraxcept in combination with nab-paclitaxel and gemcitabine in subjects with locally advanced, recurrent, or metastatic pancreatic adenocarcinoma as first line therapy. The phase 1b portion of the study is open label and patients will receive batiraxcept, nab-paclitaxel, and gemcitabine. The Phase 2 portion of the study is randomized, 2-arm, open-label study to compare efficacy and tolerability of batiraxcept, nab-paclitaxel, and gemcitabine versus nab-paclitaxel and gemcitabine as first line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Histologically or cytologically confirmed pancreatic adenocarcinoma. Must have locally advanced, recurrent, or metastatic disease ineligible for curative intent treatment(s) and eligible for first line systemic treatment.
* Must have radiologic imaging with a computed tomography (CT) scan or magnetic resonance imaging (MRI) within 22 days of study entry
* Must have at least one measurable lesion according to RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Adequate gastrointestinal (GI), bone marrow, liver and kidney function
* Life expectancy minimum of > 12 weeks
* Adequate recovery from surgery to Grade 1 or baseline with at least 28 days from time of major surgery

Exclusion Criteria:

* Received last dose of chemotherapy (neoadjuvant or adjuvant), surgery, or radiation treatment with curative intent within 6 months prior to study entry
* Islet-cell neoplasms
* Prior malignancy within the past 3 years except adequately treated basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the prostate, cervix, breast or melanoma
* Symptomatic uncontrolled central nervous system (CNS) metastasis or brain metastases unless adequately treated and controlled
* Evidence of clinically significant third spacing (e.g. pleural effusion, ascites, anasarca, etc.) within 28 days prior to study entry
* Serious active infection requiring IV antibiotics and/or hospitalization at study entry
* Active human immune deficiency (HIV) syndrome, hepatitis B, hepatitis C, or other active viral illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | 12 months
  Measured by the number of patients with AEs in Phase 1b portion of the study.
Anti-tumor activity of batiraxcept in combination with nab-paclitaxel and gemcitabine in Phase 1b portion of the study | 12 months
  Measured by Objective Response Rate (ORR): Proportion of subjects who have a partial or complete response to therapy relative to baseline in Phase 1b portion of the study.
Anti-tumor activity of batiraxcept in combination with nab-paclitaxel and gemcitabine in Phase 2 portion of the study | 30 months
  Measured by progression free survival (PFS) in patients receiving batiraxcept, nab-paclitaxel, and gemcitabine versus patients receiving nab-paclitaxel, and gemcitabine alone in Phase 2.

SECONDARY OUTCOMES:
Pharmacokinetics: AUC | 30 months
  Area under the batiraxcept concentration-time curve.
Pharmacokinetics: Cmax | 30 months
  Maximum observed batiraxcept concentration.
Pharmacokinetics: Tmax | 30 months
  Time of maximum observed batiraxcept concentration.
Pharmacokinetics: t1/2 | 30 months
  Apparent terminal half-life of batiraxcept.
Pharmacodynamic marker assessment | 30 months
  Change from the baseline in GAS6 serum levels.
Anti-drug antibody (ADA) titers | 30 months
  Change from baseline in ADA titer.
Disease control rate | 30 months
  Proportion of subjects who have a complete or partial response to therapy or maintain stable disease.
Duration of response (DOR) | 30 months
  Measured from the date of partial or complete response to therapy until the cancer progresses.
Overall survival | 60 months
  Time following the treatment until death.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - UCLA Health, Santa Monica, California
  - Boca Raton Regional Hospital / Lynn Cancer Institute, Boca Raton, Florida
  - Moffit Cancer Center, Tampa, Florida
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Michigan Medicine - University of Michigan, Ann Arbor, Michigan
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Duke University Medical Center (DUMC), Durham, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University / Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - AHN Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No